CLINICAL TRIAL: NCT00695214
Title: Drug-Induced Sleep Endoscopy for Upper Airway Evaluation in Obstructive Sleep Apnea
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other)
Responsible Party: Principal Investigator, Eric J. Kezirian, MD, MPH, Professor, Head and Neck Surgery, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-13-00379
Record Dates: First submitted 2008-06-04; First posted 2008-06-11 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; Propofol; Sleep Endoscopy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): OSA Patients considering surgical treatment
  Interventions: Drug: Propofol sedation

INTERVENTIONS:
Drug: Propofol sedation — Patients receive an intravenous propofol infusion titrated to reach a target level of sedation, sleep with arousability to verbal stimuli.

SUMMARY:
Prospective, interventional cohort study of drug-induced sleep endoscopy (DISE) to evaluate the upper airway in a cohort of obstructive sleep apnea (OSA) surgical patients. This study has investigated the reliability of this technique, demonstrating moderate-substantial interrater and test-retest reliability. This research has also compared DISE findings to those of the lateral cephalogram X-ray and examined DISE findings in individuals who have not responded to previous sleep apnea surgery. These papers have been published and available through PubMed. Additional research is ongoing, with examination of DISE findings, comparison to other evaluation techniques, and the association between DISE findings and surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with OSA considering surgical treatment

Exclusion Criteria:

* Minors
* Pregnant women
* Patients unable to provide informed consent in English themselves
* Prisoners
* Allergy to propofol, soybean oil, egg lecithin or glycerol
* Other contraindication to use of propofol (decision of anesthesiologist or otolaryngologist.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2004-02 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Association between DISE and physical examination; between DISE and polysomnogram results; between DISE and awake Mueller maneuver; between DISE and lateral cephalometry; and between DISE findings and surgical outcomes | Preoperative and postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Kezirian, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Santa Monica Medical Center, Santa Monica, California, United States

REFERENCES:
- [Background] Kezirian EJ, White DP, Malhotra A, Ma W, McCulloch CE, Goldberg AN. Interrater reliability of drug-induced sleep endoscopy. Arch Otolaryngol Head Neck Surg. 2010 Apr;136(4):393-7. doi: 10.1001/archoto.2010.26. PMID 20403857
- [Result] Rodriguez-Bruno K, Goldberg AN, McCulloch CE, Kezirian EJ. Test-retest reliability of drug-induced sleep endoscopy. Otolaryngol Head Neck Surg. 2009 May;140(5):646-51. doi: 10.1016/j.otohns.2009.01.012. PMID 19393404
- [Result] Kezirian EJ. Nonresponders to pharyngeal surgery for obstructive sleep apnea: insights from drug-induced sleep endoscopy. Laryngoscope. 2011 Jun;121(6):1320-6. doi: 10.1002/lary.21749. Epub 2011 May 6. PMID 21557231
- [Result] Kezirian EJ, Hohenhorst W, de Vries N. Drug-induced sleep endoscopy: the VOTE classification. Eur Arch Otorhinolaryngol. 2011 Aug;268(8):1233-1236. doi: 10.1007/s00405-011-1633-8. Epub 2011 May 26. PMID 21614467
- [Result] George JR, Chung S, Nielsen I, Goldberg AN, Miller A, Kezirian EJ. Comparison of drug-induced sleep endoscopy and lateral cephalometry in obstructive sleep apnea. Laryngoscope. 2012 Nov;122(11):2600-5. doi: 10.1002/lary.23561. Epub 2012 Oct 19. PMID 23086863